CLINICAL TRIAL: NCT03082001
Title: A Study to Assess the Role of Two Different Concentrations of Sucrose to Reduce Pain During Initiation of Venipuncture in Extremely Low Birth Weight Babies
Brief Title: Sucrose to Reduce Pain During Initiation of Venipuncture in Extremely Low Birth Weight Babies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELBW PAIN
Record Dates: First submitted 2017-03-02; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Neonate; Pain; ELBW
Keywords: Neonate; Pain; ELBW
MeSH Terms: conditions — Pain | interventions — Sucrose

STUDY DESIGN:
Intervention Model Description: There were two study groups A and B. The enrolled infants were administered either sterile solution of 0.2 ml of 24% sucrose or 0.2 ml of 12% sucrose 2 min prior to the procedure. The procedure involved putting first cannula in the dorm of the right hand. A 24 G needle was inserted into the vein after asepsis 2 min after the neonate had been given the allocated solution. The process was divided into three phases, the pre procedure, intraprocedure and post procedure lasting for 4 minutes. Video recording on the face of the neonate was done using a fixed video camera. The NFCS was used to evaluate and score neonatal pain.It was scored at pre, intra and post procedure 30 sec, 1 min and 2 min of the procedure.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24% Sucrose (Active Comparator): The enrolled infants were administered sterile solution of 0.2 ml of 24% sucrose (active control) 2 min prior to procedure.
  24% sucrose was prepared by mixing 2.4gm of sucrose in 10ml distilled water.
  Interventions: Drug: 24% Sucrose
- 12% Sucrose (Experimental): The enrolled infants were administered 0.2 ml of 12% sucrose 2 min prior to procedure.
  These solution were prepared under all sterile precautions by the laboratory staff unrelated to the study. 12%sucrose was prepared by mixing 1.2 gm of sucrose in 10 ml of distilled water. here were two study groups A & B. The enrolled infants were administered sterile solution of 0.2 ml of 24% sucrose (active control) 2 min prior to procedure.
  Out of these solutions 1ml was measured by 1 ml syringe and packed and covered with serially numbered opaque sealed envelopes. At the initiation of venepuncture 2 min prior to procedure 0.2 ml of solution marked with patient serial no was administered by a pre-filled syringe to the patient on the anterior aspect of the tongue avoiding spillage, by the personnel carrying out the procedure. The above mentioned personnel was blinded to the contents of the solution.
  Interventions: Drug: 12% Sucrose

INTERVENTIONS:
Drug: 12% Sucrose
  Other Names: SUGAR SOLUTION
  Arms: 12% Sucrose
Drug: 24% Sucrose
  Other Names: SUGAR SOLUTION
  Arms: 24% Sucrose

SUMMARY:
Newborn infants in the neonatal intensive care nursery experience multiple, painful tissue damaging procedures daily.

Preterm especially extremely low birth weights and critically ill newborns admitted to a Neonatal Intensive Care Unit (NICU) undergo repeated skin-breaking procedures that are necessary for their survival. Sucrose is the accepted clinical standard nonpharmacological intervention for managing acute procedural pain for these infants.

However its role in extremely low birth weight infants still need to be addressed. The exact dose and concentration of oral sucrose is still not clear.

When a Medline search was carried out to evaluate the role of two different concentrations (12% vs 24%) of oral sucrose in reducing pain in extremely low birth weight babies, very limited data was available. Cochrane Systemic Review also indicated that specific attention to the efficacy and safety of sucrose administration in extremely low birth weight preterm infants needs to be further investigated. More so, no work on this aspect was identified from the Indian subcontinent. Hence, the current study was planned with an aim to study the effects of 12% and 24% oral sucrose in extremely low birth weight infants during initiation of venipuncture and also study the side effects if any associated with these concentrations. This is a preliminary work on this topic, the results would therefore need to be interpreted with caution. However, the findings and the study design of this work will provide suitable platform for future well powered studies on this population.

DETAILED DESCRIPTION:
Research Question

• Is 0.2 ml of 12% oral sucrose not inferior to 0.2 ml of 24% oral sucrose in reducing pain during initiation of venepuncture in extremely low birth weight infants?

Research Hypothesis

• 0.2 ml of 12% oral sucrose is not inferior to 0.2 ml of 24% oral sucrose in reducing pain during initiation of venepuncture in extremely low birth weight infants.

Aims and Objective

1. To study the effect of 0.2ml of 12% & 24% oral sucrose on reducing the pain during initiation of venipuncture in Extremely Low Birth Weight (ELBW) infants.
2. To study the side effects associated with the administration of both the drugs.

Participant:

The study was conducted in the neonatal unit of Kalawati Saran Children's Hospital and Lady Hardinge Medical College, New Delhi. All the patients admitted in the neonatal units satisfying the inclusion criteria and not having any exclusion criteria were enrolled in the study.

Inclusion criteria:

* All extremely low birth weight babies (<1000gm) regardless of gestational age being admitted in NICU.
* Within first 48 hrs of post natal life
* Parental consent

Exclusion criteria:

* Neonates requiring ventilatory support.
* Neonates with any neurological impairment (HIE, seizures)
* Receiving opiates or born to mothers receiving opiates
* Newborns who have received muscle relaxants ,sedatives,analgesics
* Major congenital anomalies
* 5 mins Apgar of less than 7
* Neonates undergoing any surgery
* Birth trauma(especially precipitate deliveries)
* Instrumental delivery

Intervention

24%sucrose was prepared by mixing 2.4gm of sucrose in 10ml distilled water and 12%sucrose was prepared by mixing 1.2 gm of sucrose in 10 ml of distilled water. Out of these solutions 1ml was measured by 1 ml syringe and packed and covered with serially numbered opaque sealed envelopes. The composition of these packets were decided by a senior consultant in the department of pharmacology who had the access to the randomization sequence & was uninvolved in the study. Fresh solutions were prepared daily and unused solutions were discarded at the end of the day to be replaced with identically numbered solutions from the laboratory. All study solutions were stored in the refrigerator at 2-8°C until they were used. The patient were enrolled into the study only after an informed written consent was obtained from either of the parent / care giver. At the initiation of venepuncture 2 min prior to procedure 0.2 ml of solution marked with patient serial no was administered by a prefilled syringe to the patient on the anterior aspect of the tongue avoiding spillage, by the personnel carrying out the procedure. The above mentioned personnel was blinded to the contents of the solution.

The procedure involved putting first cannula in vein of the dorsum of right hand. Gentle steady pressure applied with the thumb to make the chosen vein prominent while the remaining fingers of the same hand helping stabilize the hand.A 24 gauge needle was inserted into vein after asepsis 2 min after the neonate had been given the allocated oral solution.The needle was inserted into vein to obtain steady blood flow.The procedure was divided into three phases. The pre-procedure phase from the beginning of the recording to just short of needle insertion. The intra-procedure phase from needle insertion to needle removal and the post-procedure phase from needle removal to end of recording lasting upto 4 min. Video recording was done by a video camera focusing on face of the patient. Neonates were monitored using a non invasive vital signs monitor to monitor their heart rate .The second video camera was focussed on the non invasive vital signs monitor.Video recording started just before oral sucrose administration and continued till 4 min after the skin puncture.All stages of needle insertion were indicated on camera by the person performing the procedure. All video recordings were evaluated independently by a consultant of the unit, who was uninvolved in the study and was blinded to the study methodology. NFCS (Neonatal facial coding system) was used to evaluate pain.The entire process involved only a single attempt at venepuncture initiation and the same was ensured rigorously during the entire study.

Sample size calculation

As there were no preliminary trials in a population of ELBW neonates comparing 12% vs 24% sucrose a convenience sample of 30 & 30 in each limb was taken.

Randomization:

Sequence Generation: Block randomization using computer generated random sequences was used with a block size of six each.

Allocation Concealment: This was done by the pharmacy which packed the 12% sucrose and the 24% sucrose into identical containers and opaque sealed envelopes sequentially labeled according to randomization code available with the consultant of Department of Pharmacology unrelated to the study.

Implementation: Randomization sequence was generated by a senior consultant in the Department of Pharmacology, unrelated to the study. The participants were enrolled for the study by the candidate according to the serial number and the candidate was blinded to the randomization code.

Blinding: The participants, the research candidate as well as the investigator assessing the painful response were blinded to the group assignment .Randomization codes and allocation sequences were broken only after the data analysis was finished.

Statistical Methods: The data was analyzed using Strata (version 11.2). Descriptive statistics (Mean, SD), Median (Range) were calculated. For comparison of Means between different groups unpaired students's t test was used. For analysis of categorical data chi-square test was used. Continuous data was also analyzed using non-parametric Ranksum (Mann-Whitney) test. Statistical significance was assumed at a P value of <0.05.

ELIGIBILITY:
Inclusion Criteria:

* All extremely low birth weight babies (<1000gm) regardless of gestational age being admitted in NICU
* Within first 48 hrs of post natal life
* Parental consent

Exclusion Criteria:

* Neonates requiring ventilatory support
* Neonates with any neurological impairment (HIE, seizures)
* Receiving opiates or born to mothers receiving opiates
* Newborns who have received muscle relaxants, sedatives,analgesics
* Major congenital anomalies
* 5 mins Apgar of less than 7
* Neonates undergoing any surgery
* Birth trauma (especially precipitate deliveries)
* Instrumental delivery

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Response to pain as assessed by Neonatal Facial Coding Score (NFCS) | The NFCS scale was scored at pre-procedure, intra-procedure (during the initiation of venepuncture). and post 30 sec, 1 min & 2 min of procedure.
  In Neonatal Facial Coding System, ten actions were monitored which included brow bulge,eye squeeze,deepening of nasolabial furrow, open lips,vertical mouth stretch, horizontal mouth stretch,cupping of tongue,chin quiver,lip pursing to form O,and tongue protrusion.Each facial action was coded as 1 for occurrence and 0 for no occurrence/absence. The final score was assigned by adding these ten parameters.Thus minimum score could be 0 and the maximum score 10 for a preterm infants

SECONDARY OUTCOMES:
Change in the heart rate from Baseline and the maximum heart rate obtained during the procedure | It was measured pre procedure to 30 sec,1 min and 2 minutes post venepuncture
  The change in the heart rate from the baseline which was measured pre procedure was recorded.It was indicated as beats/minute.
Side effects associated with the administration of sucrose in both the groups. | Any time following 30 minutes of sucrose administration
  Side effects noted were only the immediate side effects .Total number of neonates in each arm presenting with side effects would be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: VIKRAM DATTA, MD, Study Chair — Lady Hardinge Medical College

IPD SHARING:
Plan to Share IPD: Undecided